CLINICAL TRIAL: NCT00280176
Title: Phase I Study of PS-341 in Combination With 5-Fluorouracil and External Beam Radiotherapy For The Treatment Of Locally Advanced And Metastatic Rectal Cancer
Brief Title: Bortezomib, Fluorouracil, and External-Beam Radiation Therapy in Treating Patients With Stage II, Stage III, or Stage IV Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0209; CDR0000549844 (Other: PDQ number)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: recurrent rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Bortezomib; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib — 0.7mg/m2 - 1.5mg.m2 given during Weeks 1, 2, 4 and 5 on a Monday/Thursday or Tuesday/Friday schedule, up to six weeks
  Other Names: Velcade
Drug: fluorouracil — 225mg/m2 given weekly, up to 6 weeks
  Other Names: 5FU
Radiation: radiation therapy — 180 cGy, every 5 days, up to six weeks

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bortezomib and fluorouracil together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with fluorouracil and external-beam radiation therapy in treating patients with stage II, stage III, or stage IV rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bortezomib when administered in combination with fluorouracil and external beam radiotherapy as preoperative or palliative treatment in patients with stage II-IV rectal adenocarcinoma.
* Determine the dose-limiting toxicities of this regimen in these patients.

Secondary

* Determine the dose-effect relationship of bortezomib on NF-kappa B activation induced by chemoradiotherapy.
* Determine downstream events induced by NF-kappa B activation.
* Determine downstream events related to activation of p53 in response to treatment with chemoradiotherapy and bortezomib.
* Determine the rate of complete pathologic remission in patients who undergo surgical resection of their primary tumor.
* Determine the gene expression pattern of tumors by cDNA microarray analysis before and during treatment with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib.

Patients receive bortezomib IV on days 1, 4, 8, 11, 22, 25, 29, and 32 and fluorouracil IV continuously on days 2-38. Patients also undergo external beam radiotherapy 5 days a week for 5½ weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients undergo tissue biopsy at baseline and on days 1 and 2. Samples are collected and evaluated by tissue microarray analysis for NF-kappa B pathway activation; cDNA analysis, RNase protection assay, and immunohistochemistry for analysis of downstream events induced by NF-kappa B activation; and modified TdT-mediated dUTP nick-end label for analysis of apoptosis by DNA fragmentation. NF-kappa B subunits are quantified by enzyme-linked immunosorbent assay. Serum samples are collected at baseline and stored for future studies.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed diagnosis of adenocarcinoma of the rectum meeting 1 of the following clinical staging criteria:

  * T3-T4, N0, M0 (stage II disease)

    * T4 disease defined as tumor fixed on examination or involving adjacent pelvic structures, such as the sidewall, bladder, uterus, prostate, or small bowel by ultrasound or CT scan
  * Any T, N1-2, M0 (stage III disease)
  * Any T, any N, M1 (stage IV disease)
  * Recurrent disease (any prior stage)
* Candidate for local palliative therapy or curative resection of metastatic disease
* Previously treated CNS disease allowed provided it is stable for > 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Adequate nutrition
* WBC ≥ 4,000/mm³
* ANC > 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 30 mL/min
* Bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious medical or psychiatric illness that would limit study compliance or limit survival to < 2 years
* No history of refractory congestive heart failure or cardiomyopathy
* No active coronary artery disease, myocardial infarction within the past 3 months, or cerebrovascular accident within the past 3 months
* No peripheral neuropathy ≥ grade 2
* No hypersensitivity to bortezomib, boron, or mannitol

PRIOR CONCURRENT THERAPY:

* More than 1 week since prior major surgery
* More than 28 days since prior investigational agents
* Prior chemotherapy allowed
* No prior pelvic radiotherapy (for treatment of any pelvic malignancy)
* No concurrent herbal medication (excluding vitamin and mineral supplements)
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-04; Primary Completion 2008-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 weeks
Dose-limiting toxicity | 8 weeks

SECONDARY OUTCOMES:
Dose-effect relationship of bortezomib on NF-kappa B activation induced by chemoradiotherapy | 6 weeks
Downstream events induced by NF-kappa B activation | 8 weeks
Downstream events related to activation of p53 in response to treatment with chemoradiotherapy and bortezomib | 8 weeks
Rate of complete pathologic remission | 2 years
Gene expression pattern of tumors as assessed by cDNA microarray analysis pre- and post-treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee